CLINICAL TRIAL: NCT04269733
Title: Pacing-induced Cardiomyopathy - the Importance of Right Ventricular Pacing Site and Patterns of Dyssynchronous Myocardial Activation
Brief Title: Risk of Pacing-induced Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Svend Andersens Foundation (Unknown); Peacs (Unknown); Aalborg University (Other); Karl G Andersens Fond (Unknown); Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Patricia Fruelund, MD, clinical assistant, PhD student, Aalborg University Hospital
Other Study IDs: 2020-015
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Pacemaker DDD; Atrioventricular Block; Pacing-Induced Cardiomyopathy
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with a DDD-pacemaker due to high-degree AV block
  Interventions: Device: Right ventricular pacing

INTERVENTIONS:
Device: Right ventricular pacing — Right ventricular pacing from a DDD pacemaker implanted due to high-degree AV block

SUMMARY:
This study will evaluate the association between right ventricular pacing and the risk of pacing-induced cardiomyopathy.

DETAILED DESCRIPTION:
Background:

Right ventricular (RV) pacing may lead to pacing-induced cardiomyopathy (PICM) and heart failure (HF). The detrimental effects of RV pacing have been attributed to the abnormal and dyssynchronous electrical and mechanical activation of the myocardium. The activation is affected by the RV pacing site. Understanding the consequences of different RV pacing sites and the patterns of dyssynchrony may help to choose the optimal treatment for the individual patient.

Aim and objectives:

The overall aim of this project is to investigate the association between RV pacing site and the risk of PICM. Contrast enhanced cardiac computed tomography (CT) will be applied for precise localization of the RV pacing. Furthermore, investigation of the association between PICM and different mechanical and electrical myocardial activation patterns during RV pacing will be conducted using new echocardiographic and electrocardiographic methods.

Methods:

The study is designed as a retrospective cohort study with clinical follow-up. Patients with prior pacemaker implantation due to advanced atrioventricular block will be included. The study baseline is retrospective and defined as time of pacemaker implantation and follow-up is time of inclusion. Baseline data will be extracted from the Danish Pacemaker- and ICD Registry, electronic medical records (EMR) and review of echocardiographs. Follow-up data will be extracted from existing data in the EMRs as well as generated during a follow-up visit with a clinical examination. For assessment of cardiac function, RV lead position and electrical and mechanical activations patterns, the examination will include a transthoracic echocardiography, an electrocardiogram, a 3-dimensional chest photo, and a contrast-enhanced cardiac CT. Data will be analysed for differences between those who develop PICM and those who do not.

Expected outcomes and perspectives:

The hope is that this project will generate knowledge and awareness on pacemaker treatment and the risk of PICM. Understanding the pathophysiology behind PICM is key to learning how to prevent it. Accordingly, this project has the potential to contribute to improving pacemaker treatment and the quality of care for the large and still growing PM population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* De novo DDD PM implanted at Aalborg University Hospital
* PM implantation due to advanced AV block
* Duration of pacemaker treatment ≥ 1 year at time of screening
* Normal LVEF (≥50%) prior to PM implantation
* Actively attending follow-up at the PM outpatient clinic at Aalborg University Hospital after PM implantation

Exclusion Criteria:

* No written informed consent
* Baseline TTE not available or insufficient quality for assessment of LVEF
* Contraindications to a new contrast CT if no previous contrast-enhanced cardiac CT, showing RV lead position, is available
* RV pacing load < 40%.
* Deceased
* Not attending follow-up at the PM outpatient clinic at Aalborg University Hospital after PM implantation
* Device complications with removal of original implanted pacing lead > 3 months after primary implantation
* Subjects with severe ischemic heart disease and severe valvular heart disease.
* Terminal illness or unable to provide informed consent at time of screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a normal or near-normal ejection fraction prior to pacemaker implantation who received a DDD-pacemaker due to high-degree AV block ≥ 1 years prior to screening.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Pacing-induced cardiomyopathy | After ≥ 1 years of exposure to right ventricular pacing
  Time to development of PICM. PICM is defined as ≥ 10% decrease in LVEF resulting in LVEF < 50% after pacemaker implantation.

SECONDARY OUTCOMES:
Composite endpoint of new-onset heart failure | After ≥ 1 year of exposure to right ventricular pacing
  HF diagnosis and/or HF hospitalization and/or Upgrading from a DDD PM to a CRT system after pacemaker implantation.
Change in LVEF | After ≥ 1 year of exposure to right ventricular pacing
  Change in LVEF after pacemaker implantation.
New-onset atrial fibrillation and/or atrial flutter | After ≥ 1 years of exposure to right ventricular pacing
  New diagnosis of atrial fibrillation and/or atrial flutter after pacemaker implantation.
Change in LV end-diastolic volume | After ≥ 1 years of exposure to right ventricular pacing
  Change in LV end-diastolic volume after pacemaker implantation.
Change in LV end-systolic volume | After ≥ 1 years of exposure to right ventricular pacing
  Change in LV end-systolic volume after pacemaker implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No